CLINICAL TRIAL: NCT05494619
Title: A Phase III Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study to Evaluate the Efficacy, Safety, Pharmacokinetics and Pharmacodynamics of Crovalimab in Patients With Guillain-Barré Syndrome
Brief Title: A Study to Evaluate the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of Crovalimab in Participants With Guillain-Barré Syndrome (GBS)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: This study has been withdrawn due to an internal decision. The decision was not due to any safety concerns with study drug.
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Chugai Pharmaceutical Co., Ltd. (Sponsor in Taiwan and Japan) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BN43118; 2021-002968-49 (EudraCT Number)
Record Dates: First submitted 2022-08-08; First posted 2022-08-10 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Guillain-Barré Syndrome
MeSH Terms: conditions — Guillain-Barre Syndrome | interventions — gamma-Globulins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Crovalimab (Experimental): Participants will receive a single intravenous (IV) infusion of crovalimab on Day 1 based on body weight, followed by crovalimab subcutaneous (SC) injection on Days 2, 8, 15, and 22 for a total of 4 weeks. Additionally, intravenous immunoglobulin (IVIg) background therapy will be administered once a day (QD) for 5 days.
  Interventions: Drug: Crovalimab; Drug: Intravenous immunoglobulin therapy
- Placebo (Placebo Comparator): Participants will receive a single IV infusion of placebo on Day 1 based on body weight, followed by placebo SC injections on Days 2, 8, 15, and 22 for a total of 4 weeks. Additionally, IVIg background therapy will be administered QD for 5 days.
  Interventions: Drug: Placebo; Drug: Intravenous immunoglobulin therapy

INTERVENTIONS:
Drug: Crovalimab — Crovalimab will be administered at a dose of 1000 milligrams (mg) IV (for participants with body weight ≥ 40 kilograms (kg) and <100 kg) or 1500 mg IV (for participants with body weight ≥ 100 kg) on Day 1, followed by crovalimab 340 mg SC injections on Days 2, 8, 15 and 22 in all participants.
  Arms: Crovalimab
Drug: Placebo — Placebo will be administered IV on Day 1 at a dose of 1000 mg for participants with body weight ≥ 40 kg to < 100 kg, or 1500 mg for participants with body weight ≥ 100 kg. It will be administered SC on Days 2, 8, 15, and 22 at a dose 340 mg in all participants.
  Arms: Placebo
Drug: Intravenous immunoglobulin therapy — All participants will receive background therapy of IVIg at a dose of 400 milligrams/kilograms (mg/kg) QD for 5 days.

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, pharmacokinetics, and pharmacodynamics of crovalimab compared with placebo as an add-on therapy to intravenous immunoglobulin (IVIg) in participants with severe GBS.

ELIGIBILITY:
Inclusion Criteria:

* Body weight >= 40 kg at screening
* Confirmed diagnosis of GBS according to National Institute of Neurological Disorders and Stroke (NINDS) classification system
* Onset of weakness due to GBS within 2 weeks before randomization
* Able to start the first dose of blinded study drug within 2 weeks of onset of weakness
* Able to climb a flight of stairs prior to GBS
* Unable to walk independently for >=10 meters (FG >=3) with deteriorating weakness as per investigator judgment, or FG 4 or FG 5 on the GBS-DS. These criteria must be satisfied during screening.
* Undergoing or starting IVIg treatment (400 mg/kg QD for 5 days) prior to first blinded study drug administration. Participants must be able to receive the first dose of blinded study drug before the final dose of IVIg during the 5-day period of IVIg treatment.
* A record of vaccination (<=3 years) against Neisseria meningitidis, Haemophilus influenzae type B, and Streptococcus pneumonia prior to initiation of blinded study drug, in accordance with most current local guidelines as applicable for patients with complement deficiency.
* Adequate hepatic and renal function
* For female participants of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception during the treatment period and for up to 11 months after the final dose of study treatment.

Exclusion Criteria:

* Clear clinical and historical evidence of significant or disabling acute or chronic peripheral neuropathy of alternative etiology, chronic inflammatory demyelinating polyneuropathy, severe vitamin deficiency, porphyria, or diagnosis of Charcot Marie Tooth disease or other genetic neuropathy
* History of requiring a permanent aid to walk prior to GBS
* Treatment with plasmapheresis or PLEX after GBS diagnosis, or a plan to receive this treatment
* Receipt of systemic immunosuppressive treatment within 4 weeks prior to randomization
* Known or suspected hereditary complement deficiency
* Known or suspected immune deficiency
* Recent use (up to five half-lives) of treatment with complement inhibitors (e.g., 10 weeks for eculizumab, 41 weeks for ravulizumab)
* History of Neisseria meningitidis infection within 12 months prior to screening and up to first blinded study drug administration (Day 1)
* Contraindication that would prevent use of any class of antibiotics as Neisseria meningitides prophylaxis
* Immunization with a live attenuated vaccine within 1 month before first blinded study drug administration (Day 1)
* Participants who have been partially or fully vaccinated against SARS-CoV-2 with a locally approved vaccine are eligible to be enrolled in the study, 3 days or longer after inoculation.
* Recent SARS-CoV-2 infection (defined by a positive PCR test within the 2-week period prior to screening), or ongoing symptoms of active COVID-19
* Any systemic bacterial, viral, or fungal infection ongoing at screening and up to the first blinded study drug administration (Day 1) which, in the investigators' judgment, is active and could potentially be worsened by immunosuppression
* Current hepatitis B, hepatitis C, or HIV infection
* History of malignancy within 5 years prior to screening and up to the first blinded study drug administration (Day 1)
* History of hypersensitivity, allergic, or anaphylactic reactions to crovalimab or IVIg, including hypersensitivity to human, humanized, or murine monoclonal antibodies, or known hypersensitivity to any constituent of the products
* For participants with prior exposure to anti-CD20 agents, most recent anti-CD20 treatment within 6 months prior to screening
* Substance abuse within 12 months prior to screening, in the investigator's judgment
* Active suicidal ideation within 6 months prior to screening or history of suicide attempt within 3 years prior to screening
* Concurrent disease, treatment, procedure or surgery, or abnormality in clinical laboratory tests that could interfere with the conduct of the study, may pose any additional risk for the patient, or would, in the opinion of the investigator, preclude the patient's safe participation in and completion of the study
* Participation in another interventional treatment study with an investigational agent or use of any experimental therapy within 28 days of screening or within five half-lives of that investigational product, whichever is longer
* Splenectomy <= 6 months prior to screening
* Selective IgA deficiency with development of antibodies to IgA
* Only applicable for participants receiving proline-containing IVIg products: History or ongoing hyperprolinaemia type I or II at screening
* Only applicable for participants receiving sucrose/glucose/maltose-containing IVIg products: History of or ongoing diabetes mellitus or use of concomitant nephrotoxic medications
* Pregnancy or breastfeeding, or intention of becoming pregnant during the study or within 11 months after the final dose of crovalimab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-11-30 (Estimated); Primary Completion 2026-03-19 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants who Reach Hughes Functional Grade (FG) Score ≤ 1 on the Guillain-Barré Syndrome Disability Scale (GBS-DS) at Week 24 | Week 24
  The Guillain-Barré Syndrome disability score (GBS DS) is used to assess the degree of functional disability of study participants. The scale consists of seven grades of functional disability ranging from 0 (healthy with no symptoms attributable to GBS) to 6 (death).

SECONDARY OUTCOMES:
Time to Recover Independent Walking Assessed Using the 10-Meter Walk Test (10-MW) | Up to approximately 52 weeks
  Defined as time from randomization to the first time point at which the participant is able to walk independently, assessed using the 10-MWT.
Functional Outcome on GBS-DS at Week 8 | Week 8
  The Guillain-Barré Syndrome disability score (GBS DS) is used to assess the degree of functional disability of study participants. The scale consists of seven grades of functional disability ranging from 0 (healthy with no symptoms attributable to GBS) to 6 (death).
Percentage of Inflammatory Rasch-Built Overall Disability Scale (I-RODS) Responders at Week 24 | Week 24
  Defined as a participant who is able to perform all activities assessed by the I-RODS with or without some difficulties (graded 1 or 2). I-RODs is a 24-item scale to rate a participant's general ability to function and complete activities of daily living. The items range in difficulty from very easy ("reading a newspaper/book" and "eating") to very difficult ("standing for hours" and "running"). The participant assigns a score between 0 and 3 (0: not possible, 1: possible with difficulty, 2: possible without any difficulty, 3: unable to perform before GBS [option 3 only available at the baseline visit]) to each item.
Mean Post-Recovery Time | Randomization to Week 24
  Defined as the time from reaching FG ≤ 1 for the first time after randomization to Week 24
Duration of Ventilator Support | Randomization to Week 24
Percentage of Participants with Treatment Emergent Adverse Events | Up to approximately 52 weeks
  Adverse events severity was determined according to National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (NCI CTCAE v5.0) grading
Percentage of Participants with Treatment Emergent Adverse Events Leading to Study Drug Discontinuation | Up to approximately 52 weeks
Percentage of Participants with Anti-Drug Antibodies to Crovalimab | Up to approximately 52 weeks
Serum Concentrations of Crovalimab | From Day 1 up to Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm)